CLINICAL TRIAL: NCT06143566
Title: Polypill Strategy for Prevention of Cardiomyopathy Among Patients With Diabetes at Risk of Heart Failure
Brief Title: Polypill for Prevention of Cardiomyopathy
Acronym: PolyPreventHF
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ambarish Pandey, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0725
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes; High Blood Pressure
Keywords: Type 2 Diabetes; Diabetic Cardiomyopathy; Hypertension; Polypill
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Diabetic Cardiomyopathies | interventions — finerenone; empagliflozin; Losartan

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in 1:1 fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Polypill (Experimental): Participants will take a polypill containing finerenone 10 mg, empagliflozin 12.5 mg, and losartan (25, 50 mg, or 100 mg) daily.
  Interventions: Drug: Polypill
- Combined prescription of the individual medications (Active Comparator): Participants will be initiated on an SGLT2i, ARB, or finerenone if they are not already on the medication class.
  Interventions: Drug: Combined prescription of the individual medications

INTERVENTIONS:
Drug: Polypill — A combination of finerenone 10 mg, empagliflozin 12.5 mg, and losartan 50 mg or 100 mg within a polycapsule.
  Other Names: (Finerenone, Empagliflozin, Losartan)
  Arms: Polypill
Drug: Combined prescription of the individual medications — We will initiate participants on an ARB, SGLT2i, and Finerenone if they are not in the polypill arm.
  Arms: Combined prescription of the individual medications

SUMMARY:
This study will investigate the utility of a polypill-based strategy for patients with type 2 diabetes mellitus and high risk of heart failure (HF), as assessed via the WATCH-DM risk score. Polypill therapy will consist of empagliflozin 12.5 mg, losartan 25, 50 or 100 mg, and finerenone 10 mg daily. The study duration is 6 months, and participants will be randomized to either polypill therapy or simultaneous prescription of the individual drugs. The primary outcome is change in peak VO2 and adherence to usual care. The investigators hypothesize that the use of a polypill is feasible and improves medication adherence and peak VO2 as compared to those receiving usual care.

DETAILED DESCRIPTION:
Heart failure (HF) is a major cause of cardiovascular morbidity and mortality. One of the risk factors for HF is diabetes mellitus (DM). Altered glucose and lipid metabolism in DM leads to fibrosis and cardiac remodeling, ultimately causing ventricular dysfunction. While there is no consensus on the definition of "diabetic cardiomyopathy", broadly it can be defined as presence of pathological left ventricular hypertrophy, fibrosis and left ventricular diastolic/systolic dysfunction. A risk prediction score called "WATCH-DM" that includes clinical, laboratory and echocardiographic data has been developed to predict HF risk in those with type 2 DM. Every unit increase was associated with a 24% increase in relative risk of HF within 5 years. Drugs that decrease HF incidence could potentially be used in patients with Type 2 DM to alleviate HF burden. This many also improve medication adherence, which is poor for patients with polypharmacy. The rationale for the study is as follows:

* Heart failure represents a major contributor to mortality, morbidity, and healthcare costs
* Adherence to medications that prevent heart failure is low.
* A polypill strategy is an innovative approach to heart failure prevention that also promotes adherence, especially in underserved population.

The investigators propose a single-center, open-label, pragmatic, randomized study of 200 participants with T2DM and high risk of heart failure, as determined by a WATCH-DM risk score greater than or equal to 11. Duration of follow up will be 6 months. The target population is patients receiving care at UT Southwestern Medical Center or Parkland Health for Type 2 Diabetes Mellitus and high risk of heart failure. 100 participants will receive polypill and 100 will receive simultaneous individual prescriptions.The polypill will contain empagliflozin 12.5 mg, losartan 50 or 100 mg, and finerenone 10 mg and is dosed once daily. Our primary outcome will be the change in peak VO2 during a cardiopulmonary exercise test from baseline to 6 months. Secondary outcomes will include change in urine albumin creatine ratio, adherence, which will be assessed by the Morisky Medication Adherence Score - 8 (MMAS-8), pill count at baseline, 1 month and 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 DM
* History of chronic kidney disease, defined as an estimated glomerular filtration rate (eGFR) of 25 to 90 per minute per 1.73 m2 of body-surface area (stage 2 to 4 CKD) with a urinary albumin-to-creatinine ratio (with albumin measured in milligrams and creatinine measured in grams) of less than 5000
* With either a: High risk of HF as defined by High Watch-DM score (≥11) or Elevated natriuretic peptides or Diastolic dysfunction or left ventricular hypertrophy on echocardiography

Exclusion Criteria:

* eGFR < 25
* Congestive heart failure
* Hyperkalemia > 5.0
* Contraindication to any component of polypill
* Pregnancy
* Creatinine >2.0mg/dL in men and >1.8mg/dL in women
* Inability to calculate WATCH-DM score
* Inability to undergo exercise testing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Oxygen uptake during peak exercise (Peak VO2) | Baseline, 3-month, and 6-month
  The ability of a polypill to improve or prevent declines in exercise capacity as measured by changes in peak oxygen uptake at exercise will be assessed.

SECONDARY OUTCOMES:
Urine albumin to creatinine ratio | Baseline, 3 month, and 6 month
  The ratio of urinary albumin to creatinine will be measured.

OTHER OUTCOMES:
Medication Adherence | Baseline, 1 month, 3 month, and 6 month
  Assessed via the Morisky Medication Adherence Score - 8. The score ranges from 0 to 8, with 8 meaning highest adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Ambarish Pandey, MD, MSCS, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee MMY, McMurray JJV, Lorenzo-Almoros A, Kristensen SL, Sattar N, Jhund PS, Petrie MC. Diabetic cardiomyopathy. Heart. 2019 Feb;105(4):337-345. doi: 10.1136/heartjnl-2016-310342. Epub 2018 Oct 18. No abstract available. PMID 30337334
- [Background] Segar MW, Vaduganathan M, Patel KV, McGuire DK, Butler J, Fonarow GC, Basit M, Kannan V, Grodin JL, Everett B, Willett D, Berry J, Pandey A. Machine Learning to Predict the Risk of Incident Heart Failure Hospitalization Among Patients With Diabetes: The WATCH-DM Risk Score. Diabetes Care. 2019 Dec;42(12):2298-2306. doi: 10.2337/dc19-0587. Epub 2019 Sep 13. PMID 31519694
- [Background] Filippatos G, Anker SD, Agarwal R, Ruilope LM, Rossing P, Bakris GL, Tasto C, Joseph A, Kolkhof P, Lage A, Pitt B; FIGARO-DKD Investigators. Finerenone Reduces Risk of Incident Heart Failure in Patients With Chronic Kidney Disease and Type 2 Diabetes: Analyses From the FIGARO-DKD Trial. Circulation. 2022 Feb 8;145(6):437-447. doi: 10.1161/CIRCULATIONAHA.121.057983. Epub 2021 Nov 13. PMID 34775784
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978